CLINICAL TRIAL: NCT03072914
Title: Effects of Remote Ischemic Preconditioning With Postconditioning in Patients Undergoing Superficial Temporal Artery-middle Cerebral Artery (STA-MCA) Anastomosis
Brief Title: Effects of Remote Ischemic Preconditioning With Postconditioning on Neurologic Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1405/250-007
Record Dates: First submitted 2017-02-14; First posted 2017-03-07 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-03

CONDITIONS: Moyamoya Disease; Remote Ischemic Preconditioning
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): The control group has a sphygmomanometer wound around the upper arm or lower extremity and applies the same pressure, but a 3-way stopcock is installed in the middle so that no pressure is applied.
- RIPC with RIPostC group (Active Comparator): The sphygmomanometer is closed to the lower limb and the cuff is inflated and the pressure is increased by 30 mmHg higher than the systolic blood pressure of each patient for 5 minutes. The loss of the distal pulse is confirmed by Doppler in the dorsalis pedis pulse. If there is a pulse, increase the pressure until it disappears. After 5 minutes of ischemia time, the cuff is deflated to confirm that the pulse has returned and has a reperfusion time of 5 minutes. A total of 4 cycles of 5 cycles of ischemic time and 5 minutes of reperfusion time are performed. (Estimated total 40 minutes) When the skull is started to close, RIpc with RIPostC group performs RpostC and the method is the same as the above RIPC method. (Estimated total 40 minutes)
  Interventions: Procedure: RIPC with RIPostC

INTERVENTIONS:
Procedure: RIPC with RIPostC — The sphygmomanometer is closed to the lower limb and the cuff is inflated and the pressure is increased by 30 mmHg higher than the systolic blood pressure of each patient for 5 minutes. The loss of the distal pulse is confirmed by Doppler in the dorsalis pedis pulse. If there is a pulse, increase the pressure until it disappears. After 5 minutes of ischemia time, the cuff is deflated to confirm that the pulse has returned and has a reperfusion time of 5 minutes. A total of 4 cycles of 5 cycles of ischemic time and 5 minutes of reperfusion time are performed. (Estimated total 40 minutes) When the skull is started to close, RIpc with RIPostC group performs RpostC and the method is the same as the above RIPC method. (Estimated total 40 minutes)
  Arms: RIPC with RIPostC group

SUMMARY:
In the present study, we evaluated whether RIPC with RIPostC reduce the major neurocomplication in patients undergoing STA-MCA anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists
2. Adults 18 to 65 years of age
3. In patients with planned MCA-STA anastomosis under general anesthesia
4. Patients who pre-agreed to the study

Exclusion Criteria:

1. If there is a history of peripheral vascular arterial or venous disease
2. If there is a previous history of peripheral nerve disease
3. Other brain or cerebrovascular disease
4. In case of serious cardiovascular disease, pulmonary disease, kidney disease
5. Patients who do not agree with the test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Number of major adverse event | postoperative one month
  hyperperfusion syndrome, hypoperfusion, EDH, SAH, acute infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospita, Seongnam-si, Gyeonggi-do, South Korea